CLINICAL TRIAL: NCT02009189
Title: The Value of Taurolidine Lock in Long Term Parenteral Nutrition
Brief Title: Taurolidine Lock in Long Term Parenteral Nutrition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanley Dudrick's Memorial Hospital (Other)
Responsible Party: Principal Investigator, Stanislaw Klek, Assoc. Prof., Stanley Dudrick's Memorial Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Tauro-1
Record Dates: First submitted 2013-12-08; First posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Home Parenteral Nutrition; Central Venous Catheter
Keywords: home parenteral nutrition; central venous catheter
MeSH Terms: interventions — taurolidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Saline flush
  Interventions: Drug: 2% Taurolidine Lock; Drug: 1.35% Taurolidine
- 2% Taurolidine lock (Active Comparator): Catheter lock with 2% Taurolidine
  Interventions: Drug: 2% Taurolidine Lock; Drug: 1.35% Taurolidine
- 1.35% Taurolidine with citrate (Active Comparator): Catheter lock with 1.35% Taurolidine + citrate
  Interventions: Drug: 2% Taurolidine Lock; Drug: 1.35% Taurolidine

INTERVENTIONS:
Drug: 2% Taurolidine Lock — Catheter lock with 2% Taurolidine
Drug: 1.35% Taurolidine — Catheter lock with 1.35% Taurolidine + citrate

SUMMARY:
Taurolidine alone or in combination with citrate have been proposed for locking the catheter to reduce the number of catheter infections. As there is not enough evidence to give recommendations in this regard, the study tested the hipothesis that taurolidine improves the outcome of long term paretneral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* home parenteral nutrition for at least months before enrollment
* presence of central venous cathter

Exclusion Criteria:

* home nutrition < 12 months
* catheter in peripheral vein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of CVC infections | 12 months
  Number of central venous catheter infections

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw Klek, Assoc Prof, Principal Investigator — Stanley Dudrick's Memorial Hospital
Locations (1):
- Stanley Dudrick's Memorial Hospital, Skawina, Poland

REFERENCES:
- [Background] Pittiruti M, Hamilton H, Biffi R, MacFie J, Pertkiewicz M; ESPEN. ESPEN Guidelines on Parenteral Nutrition: central venous catheters (access, care, diagnosis and therapy of complications). Clin Nutr. 2009 Aug;28(4):365-77. doi: 10.1016/j.clnu.2009.03.015. Epub 2009 May 21. PMID 19464090